CLINICAL TRIAL: NCT01648335
Title: A Prospective Study of the Effect of Treatment of First Time Traumatic Shoulder Anterior Dislocation by Immobilization in External Rotation on the Incidence of Recurrent Dislocation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: beyth01-CTIL-HMO
Record Dates: First submitted 2012-07-16; First posted 2012-07-24 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Dislocation of the Shoulder
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immobilization of the shoulder in internal rotation (Active Comparator)
  Interventions: Device: Immobilization of the shoulder in internal rotation in a soft dressing called universal shoulder immobilizer (USI)
- Immobilization of the shoulder in external rotation (Experimental)
  Interventions: Device: Immobilization of the shoulder in external rotation in a soft dressing called universal shoulder immobilizer (USI)

INTERVENTIONS:
Device: Immobilization of the shoulder in external rotation in a soft dressing called universal shoulder immobilizer (USI)
  Arms: Immobilization of the shoulder in external rotation
Device: Immobilization of the shoulder in internal rotation in a soft dressing called universal shoulder immobilizer (USI)
  Arms: immobilization of the shoulder in internal rotation

SUMMARY:
Dislocation of the glenohumeral joint of the shoulder is a common orthopedic clinical problem. The majority of the dislocations are anterior (about 95%) while the rest are posterior and inferior. After reduction of the initial dislocation, the treatment's goal is to prevent recurrent dislocations. In spite of treatment, the recurrence rate is 80-90% in the population aged 18-29. There is an age-related decrease in the recurrence rate, with the only 2-3% for ages 60-70. It has been calculated that 1 in 200 soldiers in the Israeli Army between the ages of 17 and 33 suffers from recurrent shoulder dislocations [1].

The traditional treatment for primary (first-time) shoulder anterior dislocation has been immobilization of the shoulder in internal rotation in a soft dressing called universal shoulder immobilizer (USI) for 3-6 weeks. However, there is a lack of evidence-based information to demonstrate the effectiveness of this treatment. Posterior dislocations are immobilized in external rotation. Work presented previously in the Orthopaedic Research Society and more recently at the American Academy of Orthopaedic Surgeons suggests that immobilization of the shoulder after reduction of anterior dislocation is best in external rotation and not in internal rotation. MRI studies have shown that the labral tear, which is the hallmark of most traumatic anterior dislocations, is best reduced to its anatomical position when the shoulder is immobilized in external and not in internal rotation. Preliminary data indicates that immobilization in external rotation of the primary traumatic shoulder dislocations may lower the incidence of reoccurrence.

The traditional shoulder immobilizer is a generic bandage produced by several companies. In the current study, the investigators will use a USI distributed by Uriel® company (Uriel #87), which can be modified to hold the shoulder in external rotation.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18-29
* Diagnosis of anterior traumatic dislocation of the shoulder
* First time dislocation with no history of prior shoulder instability before the present episode
* Immobilization placed within 48 hours of the acute shoulder dislocation
* Subject will be in available for 2 years of follow-up
* Signed informed consent

Exclusion Criteria:

* Mechanism of injury - motor vehicle accident
* Associated fracture of tuberosities or glenoid
* Known Collagen disorder
* Additional conditions that prevent inclusion of patient according to the physician's decision

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Study Completion 2013-07

PRIMARY OUTCOMES:
• Number of recurrent dislocations within 6 months following the primary shoulder dislocation

SECONDARY OUTCOMES:
• Range of motion of the dislocated shoulder after 6 months
Supine apprehensive test after 6 months